CLINICAL TRIAL: NCT00752089
Title: Exploratory Evaluation of an Experimental Fluoride Dentifrice Formulation Using an in Situ Remineralization/Fluoride Uptake Model
Brief Title: Experimental Dentifrice Remineralization/Fluoride Uptake in an in Situ Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Z3120510
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-05

CONDITIONS: Dental Erosion
Keywords: enamel fluoride uptake; erosion; enamel remineralization
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sodium fluoride/potassium nitrate/Isopentane dentifrice (Experimental): Participants to brush their teeth for one timed minute twice daily with a gel to foam dentifrice containing active ingredients: 1450 ppm F as sodium fluoride (NaF) and 5% potassium nitrate (KNO3) and isopentane as an excipient ingredient.
  Interventions: Drug: NaF/ KNO3/isopentane Dentifrice
- NaF/KNO3 Dentifrice (Experimental): Participants to brush their teeth for one timed minute twice daily with a gel to foam dentifrice, containing as active ingredients: 1450 ppm NaF and 5% KNO3 but no isopentane.
  Interventions: Drug: NaF/KNO3 Dentifrice
- NaF Dentifrice (Active Comparator): Participants to brush their teeth for one timed minute twice daily with a dentifrice containing 1450 ppm F as NaF.
  Interventions: Drug: NaF Dentifrice
- Placebo Dentifrice (Placebo Comparator): Participants to brush their teeth for one timed minute twice daily with a fluoride free dentifrice (0 ppm F).
  Interventions: Other: Placebo Dentifrice

INTERVENTIONS:
Drug: NaF/ KNO3/isopentane Dentifrice — Experimental toothpaste
  Arms: Sodium fluoride/potassium nitrate/Isopentane dentifrice
Drug: NaF/KNO3 Dentifrice — Experimental toothpaste
  Arms: NaF/KNO3 Dentifrice
Drug: NaF Dentifrice — Active comparator
  Arms: NaF Dentifrice
Other: Placebo Dentifrice — Placebo comparator
  Arms: Placebo Dentifrice

SUMMARY:
The purpose of this study is to determine whether an experimental fluoridated dentifrice is effective in the treatment of dental caries

DETAILED DESCRIPTION:
Topical fluorides have been proven to be clinically effective in the prevention of dental caries. It is generally agreed that anti-caries effect of fluoride (F) is mainly by decreasing the rate of enamel demineralization and enhancing the rate of enamel remineralization. An in-situ Surface Micro-hardness (SMH) test is widely used to evaluate enamel demineralization and remineralization during the caries process. Determination of fluoride uptake in-situ also provides better estimation of true fluoride bioavailability of fluoride dentifrice products. In this study, an in-situ remineralization fluoride uptake model will be used to compare the efficacy of experimental dentifrice with a marketed dentifrice and placebo dentifrice. Participants wore partial dentures containing two partially demineralized enamel specimens for two weeks- 24 hours per day, except when brushing (twice daily) with test dentifrice. Following each treatment period, the enamel specimens were analyzed for SMH recovery and fluoride uptake through microdrill enamel biopsy technique.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Aged between 18 and 78
2. Fluoride: Currently living in the Indianapolis area which has a fluoridated water supply (1 ppm F) and not taking fluoride supplements for medical reasons
3. Dentures: Currently wearing a removable mandibular partial denture with sufficient room in the posterior buccal flange area to accommodate two enamel specimens (required dimensions 12 x 7 mm). Willing and capable of wearing their removable partial dentures 24 hours per day during the experimental periods
4. Dental health:Have no current active caries or periodontal disease that may compromise the study or the health of the participants and all restorations in a good state of repair
5. Salivary flow:Have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2 mL/min; gum base stimulated whole saliva flow rate ≥ 0.8 mL/min
6. Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions
7. Consent:Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
8. General Health: Good general health with (in the opinion of the investigator) no clinically significant and/or relevant abnormalities of medical history or oral examination that could interfere with participant safety during the study period

Exclusion Criteria:

1. Antibiotics:Currently taking antibiotics or have taken antibiotics in the two weeks prior to the screening visit
2. Allergy/Intolerance:Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
3. Pregnancy:Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
4. Breast-feeding:Women who are breast-feeding.
5. Clinical Study/Experimental Medication: Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit
6. Personnel:An employee of the sponsor or the study site who is directly involved in the study

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Two to three days before the start of each treatment period participants got their teeth cleaned to remove all accessible plaque and calculus, and were provided with a fluoride free dentifrice for maintaining wash-out period and standardizing the oral conditions.
Groups:
- Overall Study: This was a single-center, examiner blind, randomized, controlled, four treatment cross-over study. Participants have used each study product twice per day for two weeks and participated in each of the four treatment periods.
Period: Overall Study
Arm/Group | Overall Study
Started | 20
Received NaF/ KNO3/ 2% Isopentane | 19
Received NaF/KNO3/ 0% Isopentane | 17
Received NaF | 18
Received Placebo | 18
Completed | 14
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Protocol Deviation | 2
Not completed — Could not attend visit 9 | 1
Not completed — Not capable of wearing partial denture | 1
Not completed — Cannot continue the study | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Participants: All randomized participants who received all four treatments NaF/ KNO3/ 2% isopentane Dentifrice, NaF/KNO3/ 0% isopentane Dentifrice, NaF Dentifrice, and placebo were included in the baseline assessment.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.31 (8.226)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Micro-hardness Recovery (SMHR) of Enamel Specimens
Description: SMH test was used to assess mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents re-hardening of enamel surface. Percent SMHR was calculated from indentation values of enamel specimens at baseline (B), after intra-oral exposure (R) and after in-vitro demineralization (D) using formula: [(D-R)/ (D-B)]*100.
Time Frame: Baseline to 14 days
Population: Per-Protocol (PP) population: All randomized participants who received at least one dose of study product, had at least one post-baseline efficacy assessments and no major protocol deviations. Missing data was not imputed. Due to drop-outs, there were differences in the "n" per treatment group.
Measure: Least Squares Mean (95% Confidence Interval); unit: % SMHR
Groups:
- NaF/ KNO3/ 2% Isopentane Dentifrice: Participants brushed their teeth for one timed minute twice daily with a gel to foam dentifrice containing active ingredients: 1450 ppm F as NaF and 5% KNO3 and as an excipient ingredient: 2% isopentane.
- NaF/KNO3/ 0% Isopentane Dentifrice: Participants brushed their teeth for one timed minute twice daily with a gel to foam dentifrice, containing as active ingredients: 1450 ppm NaF and 5% KNO3 but no isopentane.
- NaF Dentifrice: Participants brushed their teeth for one timed minute twice daily with a dentifrice containing 1450 ppm F as NaF.
- Placebo Dentifrice: Participants brushed their teeth for one timed minute twice daily with a fluoride free dentifrice (0 ppm F).
Arm/Group | NaF/ KNO3/ 2% Isopentane Dentifrice | NaF/KNO3/ 0% Isopentane Dentifrice | NaF Dentifrice | Placebo Dentifrice
Number analyzed (Participants) | 17 | 17 | 17 | 18
% SMHR | 39.46 (4.10) [31.17 to 47.75] | 38.31 (4.11) [30.00 to 46.62] | 36.17 (4.10) [27.89 to 44.44] | 17.26 (4.04) [9.08 to 25.43]
Statistical Analysis 1: Comparison: NaF/ KNO3/ 2% Isopentane Dentifrice vs NaF/KNO3/ 0% Isopentane Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.7756, ANOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = 1.146, 95% CI 2-sided [-6.904 to 9.196] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: NaF/ KNO3/ 2% Isopentane Dentifrice vs NaF Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.4194, ANOVA — No adjustments for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = 3.291, 95% CI 2-sided [-4.840 to 11.421] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF/ KNO3/ 2% Isopentane Dentifrice vs Placebo Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = 22.200, 95% CI 2-sided [14.280 to 30.120] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaF/KNO3/ 0% Isopentane Dentifrice vs NaF Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.5927, ANOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = 2.145, 95% CI 2-sided [-5.874 to 10.164] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaF/KNO3/ 0% Isopentane Dentifrice vs Placebo Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = 21.054, 95% CI 2-sided [13.189 to 28.919] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: NaF Dentifrice vs Placebo Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = 18.909, 95% CI 2-sided [11.036 to 26.783] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Adjusted Mean Change From Baseline in Enamel Fluoride Uptake
Description: Enamel fluoride uptake was determined using the microdrill enamel biopsy technique. The amount of fluoride uptake by enamel was calculated based on the amount of fluoride (F) divided by the area of the enamel cores and expressed as ug*F/cm^3. The difference between treatments was calculated with respect to fluoride uptake by enamel.
Time Frame: Baseline to 14 days
Population: PP population: All randomized participants who received at least one dose of study product, had at least one post-baseline efficacy assessments and no major protocol deviations. Missing data was not imputed. Due to drop-outs, there were differences in the "n" per treatment group.
Measure: Least Squares Mean (95% Confidence Interval); unit: ug*F/cm^3
Groups:
- NaF/ KNO3/ 0% Isopentane Dentifrice: Participants brushed their teeth for one timed minute twice daily with a gel to foam dentifrice, containing as active ingredients: 1450 ppm NaF and 5% KNO3 but no isopentane.
Arm/Group | NaF/ KNO3/ 2% Isopentane Dentifrice | NaF/ KNO3/ 0% Isopentane Dentifrice | NaF Dentifrice | Placebo Dentifrice
Number analyzed (Participants) | 17 | 17 | 17 | 18
ug*F/cm^3 | 2445.86 (256.55) [1926.90 to 2694.82] | 2767.30 (257.16) [2247.10 to 3287.50] | 2518.54 (256.55) [2000.28 to 3036.80] | 661.18 (252.88) [148.91 to 1173.46]
Statistical Analysis 1: Comparison: NaF/ KNO3/ 2% Isopentane Dentifrice vs NaF/ KNO3/ 0% Isopentane Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.1990, ANOVA — No adjustments for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = -321.438, 95% CI 2-sided [-818.118 to 175.242] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF/ KNO3/ 2% Isopentane Dentifrice vs NaF Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.7718, ANOVA — No adjustments for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = -72.680, 95% CI [-574.398 to 429.039] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF/ KNO3/ 2% Isopentane Dentifrice vs Placebo Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = 1784.675, 95% CI [1296.044 to 2273.306] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaF/ KNO3/ 0% Isopentane Dentifrice vs NaF Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.3164, ANOVA — No adjustments for multiple comparisons were made as the primary comparison was pre-defined; The model included tratment and period as fixed and participant as random factors; Adjusted mean difference = 248.758, 95% CI [-245.962 to 743.478] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaF/ KNO3/ 0% Isopentane Dentifrice vs Placebo Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period as fixed and participant as random factors; Adjusted mean difference = 2106.113, 95% CI 2-sided [1620.906 to 2591.320] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: NaF Dentifrice vs Placebo Dentifrice; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment and period and fixed and participant as random factors; Adjusted mean difference = 1857.355, 95% CI 2-sided [1371.637 to 2343.072] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 13 weeks
Groups:
- NaF/ KNO3/ 2 % Isopentane Dentifrice: Participants brushed their teeth for one timed minute twice daily with a gel to foam dentifrice containing active ingredients: 1450 ppm F as NaF and 5% KNO3 and as an excipient ingredient: 2% isopentane.
Arm/Group | NaF/ KNO3/ 2 % Isopentane Dentifrice | NaF/KNO3/ 0% Isopentane Dentifrice | NaF Dentifrice | Placebo Dentifrice
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/17 | 3/17 | 4/18 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF/ KNO3/ 2 % Isopentane Dentifrice (N=17) | NaF/KNO3/ 0% Isopentane Dentifrice (N=17) | NaF Dentifrice (N=18) | Placebo Dentifrice (N=18)
Gingival erythema (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No